CLINICAL TRIAL: NCT02867280
Title: A Prospective Multicenter Non-randomized Controlled Study of Sorafenib (Nexavar) Treatment in Patients With Hepatocellular Carcinoma With Microvascular Invasion After Radical Resection
Brief Title: Sorafenib Treatment in Patients With Hepatocellular Carcinoma With Microvascular Invasion After Radical Resection
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Midterm analysis showed negative results.
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Chen Min-Shan, Director of the Department of Hepatobiliary Surgery, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sorafenib-MVI
Record Dates: First submitted 2016-07-10; First posted 2016-08-15 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Hepatocellular Carcinoma; Recurrence
Keywords: Sorafenib; Microvascular invasion; adjuvant therapy; hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sorafenib (Experimental): Sorafenib (Nexavar) 200mg tablet, 2 tablets oral daily for 2 years, starting within 4weeks after hepatectomy. Regular treatment combined.
  Interventions: Drug: Sorafenib
- Control (No Intervention): No use of Sorafenib (Nexavar). Regular treatment.

INTERVENTIONS:
Drug: Sorafenib — red round tablet
  Other Names: Nexavar
  Arms: Sorafenib

SUMMARY:
This prospective multicenter non-randomized controlled study evaluates the efficacy and safety of treatment with Sorafenib (Nevaxar) in patients with hepatocellular carcinoma with microvascular invasion after radical resection compared to conventional therapies.

DETAILED DESCRIPTION:
The study is a multicenter, non-randomized, open-label, blank controlled study which initiated by Investigators. The study population include patients without macroscopic vascular invasion and distant metastasis, undergoing R0 resection, postoperative pathology confirming hepatocellular carcinoma with microvascular invasion (MVI) (BCLC A or B stage; T2 or part T3aN0M0). The primary end point of this study is recurrence free survival（RFS）at the 2nd postoperative years, and the secondary end points include postoperative median time to recurrence (TTR), 1-year, 3-years, 5-years postoperative recurrence free survival (RFS), 3-years, 5-years postoperative overall survival, and safety and tolerance of sorafenib as an adjuvant therapy for HCC. Patients in the treatment group will start Sorafenib within 4 weeks after hepatectomy at doze of 400mg per day, and last continuously for 2 years, or until disease progression. Patients in the control group will take regular treatment with no use of Sorafenib. Both groups are forbid receiving postoperative anti-cancer therapy such as adjuvant radiotherapy, chemotherapy and TACE. Patients of both groups should receive antiviral therapy according to guidelines. Chinese traditional medicine and nutritional support can be used without limitation, and the information of concomitant drug need to be recorded for further analysis. Treatment for relieve drug related AEs can be used as needed. Patients of both groups will be treated with best clinical practice as routine after confirmed recurrence/metastasis, and the information of further treatment need to be recorded and follow-up till death.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years
2. Hepatocellular carcinoma confirmed by pathology
3. No macroscopic tumor thrombus vascular invasion and distant metastasis
4. R0 resection（clean resection margin both macroscopically and microscopically）
5. MVI confirmed by pathology
6. ECOG 0-1
7. Child-Pugh stage A
8. WBC > 3×10E9/L；HB > 90 G/L；PLT > 50×10E9/L
9. ALT，AST not exceeding 5 times of the upper limit of normal value；CRE，TBIL not exceeding 1.5 times of the upper limit of normal value

Exclusion Criteria:

1. Tumor rupture or invading to adjacent organs
2. Patients who underwent liver transplantation
3. Past history of or simultaneously receiving other anti-cancer therapy (such as TACE, chemotherapy, radiotherapy and others）and immune cell infusion therapy
4. Uncontrolled cardiovascular and cerebrovascular diseases
5. History of gastrointestinal bleeding within 6 months
6. Active infection other than HBV, HCV
7. Postoperative complications, not suitable to take Sorafenib (such as long term use of drainage due to bile leakage, poor wound healing and others)
8. Confirmed liver cancer recurrence or metastasis within 4 weeks after hepatectomy
9. Poor compliance, cannot adhere to regular follow up
10. Diagnosed with other original malignant tumors other than HCC

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Recurrence free survival | 2 years
  To determine the recurrence free survival rate at 2 years after hepatectomy

SECONDARY OUTCOMES:
Time To Recurrence | From date of liver resection until the date of first documented relapse, assessed up to 5 years
  To determine the median postoperative time to recurrence
Recurrence rate | 2 years
  To determine the recurrence rate within 2 years after hepatectomy
Recurrence free survival | 1year, 3years, 5 years
  To determine the recurrence free survival at postoperative 1-year, 3-year, and 5-year
Overall survival | 3 years, 5 years
  To determine the overall survival at postoperative 3-year and 5-year
Incidence of Treatment-related Adverse Events measures using CTCAE v4.0 | 2 years
  measures using CTCAE v4.0
Incidence of dose modification of sorafenib due to adverse events. | 2 years
  The actual total dose of sorafenib for every patients will be collected as well.

CONTACTS AND LOCATIONS:
Overall Officials: Minshan Chen, PHD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No